CLINICAL TRIAL: NCT00639808
Title: Multicenter, Randomized, Double-Blind, Placebo Controlled, Crossover Single Dose Study to Assess Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Effect on Gastric Emptying of TZP-101 IV Infusion in Diabetic Gastroparesis Patients
Brief Title: Safety and Efficacy of IV Infusion of Investigational Agent (TZP-101) in Patients With Diabetic Gastroparesis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tranzyme, Inc. (Industry)
Responsible Party: Gordana Kosutic, MD; VP Clinical & Regulatory Affairs, Tranzyme, Inc.
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TZP-101-CL-002; EudraCT 2006-002730-38
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2008-03-20 (Estimated); Status verified 2008-03

CONDITIONS: Gastroparesis; Diabetes Mellitus
Keywords: delayed gastric emptying; symptomatic gastroparesis; diabetes mellitus
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Glucose; Water; ulimorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: 5% dextrose in water
- 2 (Experimental): TZP-101
  Interventions: Drug: TZP-101

INTERVENTIONS:
Drug: 5% dextrose in water — 60 ml IV infusion over 30 minutes
  Other Names: D5W
  Arms: 1
Drug: TZP-101 — 1 infusion: IV 2ml/min for 30 minutes for 1 day of either 160, 320 or 600 micrograms/kg
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether TZP-101 is safe in people with diabetes. Also to determine if TZP-101 is effective in increasing the gastric emptying rate in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject has type 1 or type 2 diabetes mellitus
* Subject has documented diagnosis of gastroparesis by:
* Delayed gastric emptying (gastric retention ≥60% at 2h and ≥10% at 4 h; based on scintigraphy -4h standardized radionuclide solid meal)
* A minimum 3 month history of chronic upper abdominal discomfort (two or more: chronic postprandial fullness, bloating, epigastric discomfort, early satiety, belching after meal, postprandial nausea, vomiting)
* Subject has normal upper endoscopy
* If female, must be permanently sterilized or postmenopausa.

Exclusion Criteria:

* Patient has received any investigational drug within the preceding 30 days
* Patient is taking unstable doses of medication that affects gastric motility
* Patient has co-morbid condition
* Patient has a positive laboratory test result for hepatitis B, hepatitis C, HIV, or controlled substances.
* Patient has a history of a psychiatric disorder (including drug or alcohol addiction) requiring care by a psychiatrist or psychologist within the preceding 12 months.
* Patient has a recent,adult history of clinically significanthypersensitivity reaction(s) to any drug.
* Patient has known history of alcoholism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
12-lead ECG data | 8 assessments including baseline (prior to start of infusion of study drug) until 24 four hours after start of infusion.

SECONDARY OUTCOMES:
Scintigraphy to measure rate of gastric emptying after ingestion of a radio-labeled meal | Measurements at: 30, 60, 120, 180, 210, and 240 minutes after the meal is eaten

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (2):
  - Aarhus Hospital, Aarhus
  - Hvidore Hospital, Copenhagen
- Karolinska University Hospital, Stockholm, Sweden